CLINICAL TRIAL: NCT00847223
Title: A Phase II Study Evaluating the Efficacy and Safety of the Farnesyl-transferase Inhibitor ZARNESTRA® in Patients With Relapsed, Refractory or Progressive Mantle Cell Lymphoma Not Appropriate for Autologous Bone Marrow Transplantation
Brief Title: Efficacy and Safety of the Farnesyl-transferase Inhibitor (Tipifarnib) in Mantle Cell Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inefficiency of treatment
Sponsor: Lymphoma Study Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCL06-1
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Mantle Cell Lymphoma
Keywords: Mantle cell lymphoma; Lymphoma; relapsed, refractory or progressive MCL; Mantle cell lymphoma (relapsed, refractory or progressive)
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma; Recurrence | interventions — tipifarnib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ZARNESTRA (Tipifarnib) (Experimental)
  Interventions: Drug: ZARNESTRA (Tipifarnib)

INTERVENTIONS:
Drug: ZARNESTRA (Tipifarnib)

SUMMARY:
To determine the EFFICACY and the SAFETY PROFILE and TOXICITY of Zarnestra® in the treatment of patients with previously treated mantle cell lymphoma not appropriate for autologous bone marrow transplantation. 27 evaluable subjects will be enrolled for an analysis in 2 stages (11 for the first stage, 16 for the second).

Patients who receive at least one dose of Zarnestra® and have at least one post-baseline response assessment of discontinued study frug for early progression are evaluable. Subjects not evaluable for response will be replaced, up to 35 patients.

DETAILED DESCRIPTION:
Zarnestra® will be administered at 300 mg administered orally twice daily for the first 21 days of each 28-days cycle. Tipifarnib treatment stops no later than day 21 of each cycle.

Subjects will receive a total of 4 cycles of treatment. Two additional cycles might be administered for patients showing improvement to PR after 4 cycles.

After testing the drug on 11 patients in the first stage, the trial will be terminated if 1 or fewer respond and the drug will not be considered as effective.

If two or more patients respond in the first stage, the trial goes on to the second stage to include a total of 27 patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject 18 years or older.
* Initial diagnosis of histologically confirmed mantle cell lymphoma based on the World Health Organization 1997 classification.
* Patient not able to receive high dose autologous stem cell transplantation with relapsed, refractory or progressive MCL after prior anti-neoplastic treatment. Relapse or progression since previous anti-neoplastic therapy must be documented by new lesions or objective evidence of progression of existing lesions. Biopsy is not required.
* Ann Arbor stages I-IV.
* At least 1 measurable lymph node mass that is >1.5 cm in 2 perpendicular dimensions, and has not been previously irradiated or has grown since previous irradiation.
* Eastern Cooperative Oncology Group [ECOG] performance status 0-2.
* The following laboratory values at screening,:

  * Absolute neutrophil count (ANC) ≥ 1.0 G/L and Platelets ≥ 75 G/L
  * Aspartate transaminase (AST) ≤ 2.5 x ULN; Alanine transaminase (ALT) ≤ 2.5 x ULN; Total bilirubin ≤ 1.5 x ULN; Creatinin level ≤ 150 µmol/L
* Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (ie, a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study. Women are neither breast feeding nor pregnant for the duration of the study. Confirmation that the subject is not pregnant must be established by a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women. Male subject agrees to use an acceptable method for contraception for the duration of the study.
* Voluntary signed informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Patient with minimum life expectancy of 3 months.

Exclusion Criteria:

* Any other type of lymphoma.
* Previous treatment with Zarnestra®.
* Anti-neoplastic or radiation therapy within 2 weeks before Day 1 of Cycle 1.
* Major surgery within 2 weeks before Day 1 of Cycle 1.
* Rituximab, alemtuzumab (Mabcampath®), or other unconjugated therapeutic antibody within 2 weeks before Day 1 of Cycle 1
* Nitrosoureas within 2 weeks before Day 1 of Cycle 1.
* Radioimmunoconjugates or toxin immunoconjugates such as ibritumomab tiuxetan (Zevalin™), or tositumomab (Bexxar®) within 4 weeks before Day 1 of Cycle 1.
* Less than 30 days since participation in another investigational agent study on Day 1 of cycle 1. Concurrent participation in non-treatment studies is allowed, if it will not interfere with participation in this study.
* Known or suspected allergy to imidazole drugs, such as clotrimazole, ketoconazole, miconazole, econazole, fenticonazole, isoconazole, sulconazole, tioconazole, or terconazole.
* Subjects not adequately recovered from any treatment-related non hematologic toxicity (recovery is defined as NCI CTC v3.0 Grade 0 or 1).
* Symptomatic peripheral neuropathy of any grade.
* Diagnosed or treated for a malignancy other than NHL within 5 years before Day 1 of Cycle 1, with the exception of complete resection of basal cell carcinoma, squamous cell carcinoma of the skin, or in situ malignancy. Subjects previously diagnosed with prostate cancer are eligible if (1) their disease was T1-T2a, N0, M0, with a Gleason score ≤7, and a prostate specific antigen (PSA) ≤10 ng/mL prior to initial therapy, (2) they had definitive curative therapy (ie, prostatectomy or radiotherapy) ≥2 years before Day 1 of Cycle 1, and (3) at a minimum 2 years following therapy they had no clinical evidence of prostate cancer, and their PSA was undetectable if they underwent prostatectomy or <1 ng/mL if they did not undergo prostatectomy.
* Active systemic infection requiring treatment.
* Previously known HIV positive serology
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Adult patient under guardian.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-06 (Actual); Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Overall response rate (complete response [CR] + complete response unconfirmed [CRu] + partial response [PR]) | 4 months
  Percentage of patients in CR, CR uncertain or PR

SECONDARY OUTCOMES:
Overall CR rate (CR + CRu) | 2 years
  percentage of patients in CR or CRu
Progression-free survival (PFS) | 2 years
  duration of survival without progression
overall survival | 2 years
  percentage of patients alive
number of SAE | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Catherine THIEBLEMONT, MD, Study Chair — Lymphoma Study Association; Hervé TILLY, MD, Principal Investigator — Lymphoma Study Association; Catherine SEBBAN, MD, Principal Investigator — Lymphoma Study Association; Bertrand COIFFIER, MD, Principal Investigator — Lymphoma Study Association; Serge BOLOGNA, MD, Principal Investigator — Lymphoma Study Association; Olivier CASASNOVAS, MD, Principal Investigator — Lymphoma Study Association; Richard DELARUE, MD, Principal Investigator — Lymphoma Study Association; Réda BOUABDALLAH, MD, Principal Investigator — Dr; Franck MORSCHHAUSER, MD, Principal Investigator — Lymphoma Study Association